CLINICAL TRIAL: NCT07334041
Title: Comparison of Preoxygenation Techniques in Healthy Volunteers With Monitoring of End-tidal Oxygen Fraction (FeO₂) and Oxygen Reserve Index (ORI).
Acronym: OXYGAME1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHUO-2025-21
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Preoxygenation; High flow nasal cannula; Non-invasive ventilation; Healthy volunteers; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Randomized interventional crossover study comparing two preoxygenation techniques in healthy volunteers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive ventilation combined to high flow nasal cannula (Experimental): - NIV + HFNC: Non-invasive ventilation in pressure-controlled mode with inspiratory pressure adjusted to achieve a tidal volume of 6-8 mL/kg (in practice, inspiratory pressure between 5 and 10 cmH₂O) and a PEEP of 5 cmH₂O, combined with high-flow nasal cannula oxygen at 60 L/min with an FiO₂ of 100%
  Interventions: Other: Preoxygenation with VNI + OHD
- Non invasive ventilation (Experimental): - NIV alone in pressure-controlled mode with inspiratory pressure adjusted to achieve a tidal volume of 6-8 mL/kg (in practice, inspiratory pressure between 5 and 10 cmH₂O) and a PEEP of 5 cmH₂O
  Interventions: Other: Preoxygenation with VNI

INTERVENTIONS:
Other: Preoxygenation with VNI + OHD — Each preoxygenation session will last 3 minutes with the participant positioned at a 30° head-up angle.
  A washout period of 10 minutes will be applied between each preoxygenation session, and initiation of the second preoxygenation technique will require the Oxygen Reserve Index (ORI) to return to 0.
  Monitoring will include:
  * Oxygen Reserve Index (ORI)
  * End-tidal oxygen fraction (FeO₂) measured at the NIV mask
  * Peripheral oxygen saturation (SpO₂)
  Arms: Non-invasive ventilation combined to high flow nasal cannula
Other: Preoxygenation with VNI — Each preoxygenation session will last 3 minutes with the participant positioned at a 30° head-up angle.
  A washout period of 10 minutes will be applied between each preoxygenation session, and initiation of the second preoxygenation technique will require the Oxygen Reserve Index (ORI) to return to 0.
  Monitoring will include:
  * Oxygen Reserve Index (ORI)
  * End-tidal oxygen fraction (FeO₂) measured at the NIV mask
  * Peripheral oxygen saturation (SpO₂)
  Arms: Non invasive ventilation

SUMMARY:
The objective of this physiological study is to compare two preoxygenation techniques (non-invasive ventilation combined with high-flow nasal oxygen versus non-invasive ventilation alone) by monitoring end-tidal oxygen fraction (FeO₂) and the Oxygen Reserve Index (ORI) during 3 minutes of preoxygenation in healthy volunteers.

DETAILED DESCRIPTION:
An intubation procedure is performed in several successive phases:

1. Preoxygenation phase: This phase consists of administering 100% oxygen for 3 to 5 minutes in order to increase oxygen reserves.
2. Alveolar hypoventilation phase: This phase begins with the administration of anesthetic agents, leading to a reduction in spontaneous ventilation.
3. Apnea phase: During this phase, laryngoscopy is performed and the endotracheal tube is inserted into the trachea.
4. Initiation of invasive mechanical ventilation: Once intubation is successful, the patient is placed on assisted mechanical ventilation.

Several devices can be used to perform preoxygenation:

* Bag-valve mask (BVM)
* High-flow nasal cannula therapy (HFNC)
* Non-invasive ventilation (NIV):

Current recommendations from critical care societies suggest the use of:

* BVM or HFNC for non-hypoxemic patients
* NIV for hypoxemic patients A single-center randomized controlled study (OPTINIV) demonstrated the benefit of combining NIV and HFNC for preoxygenation. However, placing an NIV mask over HFNC nasal cannulae may result in mask leaks, leading to ambient air entrainment, as well as a potential risk of excessive airway pressure related to HFNC. In this study, HFNC cannulae in the control group were left in place but inactive. Consequently, it remains difficult to determine whether the observed efficacy of the NIV + HFNC combination was related to leak compensation by HFNC during preoxygenation, or to apneic oxygenation provided by HFNC between laryngoscopy and successful intubation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Healthy volunteer who has provided written informed consent
* Age > 18 years

Exclusion Criteria:

* Long-term oxygen therapy
* Cardiac or pulmonary disease (including asthma)
* Presence of Raynaud's syndrome
* Claustrophobia
* Body mass index (BMI) ≥ 30 kg/m²
* Presence of nail polish preventing accurate SpO₂ and ORI measurement
* Under legal protection
* Incarcerated individuals
* Persons deprived of liberty
* Not affiliated to French social security
* Pregnant or breastfeeding women
* Individuals currently participating in a drug study and still within the exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in end-tidal oxygen fraction (FeO2) at the end of each preoxygenation technique | 3 minutes
  FeO2 will be collected every 12 seconds during preoxygenation. The mean FeO2 value at 3 minutes will be used for comparison between techniques.

SECONDARY OUTCOMES:
Change in end-tidal oxygen fraction (FeO2) during each preoxygenation technique | 3 minutes
  Change in end-tidal oxygen fraction (FeO₂) will be evaluated by recording FeO₂ every 12 seconds during the 3-minute preoxygenation period.
Maximum FeO2 value | 3 minutes
  Maximum FeO2 value achieved during the 3 minutes of each preoxygenation technique
Average Oxygen Reserve Index (ORI) value | 3 minutes
  The ORI will be recorded every 30 seconds during preoxygenation. The mean ORI value at 3 minutes will be used for comparison.
Maximum ORI value | 3 minutes
  Maximum ORI value achieved during the 3 minutes of each preoxygenation technique
Change in ORI during each preoxygenation technique | 3 minutes
  Change in ORI will be evaluated by recording ORI every 2 seconds during the 3 minutes of preoxygenation.
Time (in seconds) required to reach an ORI value ≥ 0.60 and FeO2 ≥ 90% during the 3 minutes of each preoxygenation technique | 3 minutes
Time (in seconds) for ORI to return to 0 after cessation of preoxygenation. | 3 minutes
Change in peripheral oxygen saturation (SpO2) during each preoxygenation technique | 3 minutes
  The change in SpO2 will be evaluated by recording SpO2 every 12 seconds during the 3 minutes of preoxygenation.
Change in ventilator parameters (inspiratory and expiratory tidal volumes) | 3 minutes
  Change in inspiratory and expiratory tidal volumes measured every 30 seconds during the 3 minutes of preoxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAH, MD, Principal Investigator — CHU d'Orléans
Locations (1):
- CHU Orléans, Orléans, France